CLINICAL TRIAL: NCT04297176
Title: Clinical and Economic Evaluation of Optimal Monitoring Parameters and Sampling Schemes for Vancomycin Therapeutic Drug Monitoring in Qatar
Brief Title: Economic Evaluation of Vancomycin Therapeutic Drug Monitoring Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Qatar University (Other)
Responsible Party: Principal Investigator, Dr. Eman Zeyad Ibrahim Elmekaty, Clinical Pharmacist, Infectious Diseases Department, Communicable Diseases Center, Study Principle Investigator, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15418/15
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Infection, Bacterial
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional monitoring method (Experimental): Patients are dosed using two timed vancomycin serum concentrations
  Interventions: Drug: Vancomycin-traditional dosing
- One concentration method (Active Comparator): Patients are dosed based on one timed vancomycin serum level
  Interventions: Drug: Vancomycin- Trough-only based dosing

INTERVENTIONS:
Drug: Vancomycin-traditional dosing — The dose is calculated based on 2 vancomycin serum levels
  Arms: Traditional monitoring method
Drug: Vancomycin- Trough-only based dosing — The dose is calculated based on 1 vancomycin serum level (i.e. trough)
  Arms: One concentration method

SUMMARY:
Vancomycin is a widely used antibiotic in the treatment of complicated gram positive infections. Approaches to vancomycin therapeutic drug monitioring (TDM) vary. This clinical trial aimed to compare the pharmacoeconomic outcomes between various vancomyicn TDM approaches.

Research questions: Which vancomycin therapeutic drug monitoring (TDM) approach is associated with superior economic outcomes?

-Objectives: In this proposed multicenter randomized controlled trial (RCT), we aim to compare the pharmacoeconomic outcomes of various vancomycin TDM approaches.

ELIGIBILITY:
Inclusion Criteria:

* adults at least 18 yrs who are hospitalized and initiated on IV vancomycin

Exclusion Criteria:

* renal instability
* immunosuppression;
* vancomycin allergy;
* history of recurrent peritonitis
* administration of < 4 doses of vancomycin
* pregnancy;
* hemoglobin < 8 g/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
therapeutic success | The follow up time varies according to the infection type. It ranges from 7 days to 1 month.
  Therapeutic success will be assessed as therapeutic cure (composite endpoint)or therapeutic failure (composite endpoint). Therapeutic cure is defined as clinical cure and/or microbiologic cure . Clinical cure is defined as the absence of infection signs/symptoms without the need for additional antibiotic treatment. Microbiologic cure is defined as negative blood cultures at 5 days after vancomycin treatment initiation. Therapeutic failure includes at least one of the following -clinical failure, microbiologic failure, premature discontinuation due to ADR or all-cause mortality. Clinical failure is defined as insufficient clinical response to initial vancomycin therapy necessitating antibiotic change. Microbiological failure is defined as a positive culture at ≥ 5 days after initiation of vancomycin treatment.
cost-benefit | Ranges from 7 days to 1 month, according to the infection type and possible antibiotic changes if treatment failure occurs
  The hospital and treatment related costs will be compared between the two study arms, from a hospital perspective, associating the clinical outcomes mentioned in Outcome 1 above. The arm showing least costs will be determined as more beneficial to the healthcare system.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No